CLINICAL TRIAL: NCT07064187
Title: Evaluate The Improvement In Symptoms Of Patients Using Cationorm After Pterygium Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nguyen Viet Giap (Other)
Responsible Party: Sponsor-Investigator, Nguyen Viet Giap, Director of Hospital, Ba Ria - Vung Tau Eye Hospital
Organization: Ba Ria - Vung Tau Eye Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 30/BVM-KHTH No.2
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Ocular Discomfort
Keywords: cationorm; artificial tear; pterygium surgery
MeSH Terms: interventions — Cationorm; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cationorm arm (Experimental): Participants will take:
  * Before surgery: 1 drop Cationorm at the eye that will undergo surgery
  * After surgery: 1 drop Cationorm at the eye that underwent surgery before eye bandages
  * Follow up after surgery: 1 drop Cationorm 4-6 times/day alternating with antibiotics (third-fourth generation quinolone) with 2-hour interval between drops
  * Maintenance phase: 7-14 days with the same regimen
  Interventions: Drug: Cationorm single-dose eye drop
- Artificial tear arm (Active Comparator): Participants will take:
  * Before surgery: 1 drop artificial tear at the eye that will undergo surgery
  * After surgery: 1 drop artificial tear at the eye that underwent surgery before eye bandages
  * Follow up after surgery: 1 drop artificial tear 4-6 times/day alternating with antibiotics (third-fourth generation quinolone) with 2-hour interval between drops
  * Maintenance phase: 7-14 days with the same regimen
  Interventions: Drug: Artificial tear eye drop

INTERVENTIONS:
Drug: Cationorm single-dose eye drop — Cationorm single-dose eye drop is a preservative-free, cationic oil-in-water nano-emulsion.
  Other Names: Cationic emulsion
  Arms: Cationorm arm
Drug: Artificial tear eye drop — Artificial tear eye drops are hyaluronic acid, polymers or cellulose derivatives eye drops
  Arms: Artificial tear arm

SUMMARY:
The goal of this interventional clinical trial is to learn whether Cationorm can improve symptoms after pterygium surgery. The main question it aims to answer is what is the level of improvement of symptoms after pterygium surgery.

Researchers will compare with other artificial tears (hyaluronic acid, polymers or cellulose derivatives eye drops) arm to see if Cationorm is similar or superior in terms of improvement of symptoms after pterygium surgery.

Participants will

* Take 1 drop Cationorm/artificial tear before and after surgery and during follow up.
* Visit for checkups after 7 days

DETAILED DESCRIPTION:
Participants will take:

* Before surgery: 1 drop Cationorm/artificial tear at the eye that will undergo surgery
* After surgery: 1 drop Cationorm/artificial tear at the eye that underwent surgery before eye bandages
* Follow up after surgery: 1 drop Cationorm/artificial tear 4-6 times/day alternating with antibiotics (third-fourth generation quinolone) with 2-hour interval between drops
* Maintenance phase: 7-14 days with the same regimen
* After day 5, if fluorescein staining (-), can add corticosteroid monotherapy or addition with antibiotics
* After 5 days of surgery, can add more antibiotics depend on the symptoms of patients

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-70 years
* Having diagnosis of pterygium grade II or III and planning for pterygium surgery
* Giving consent to participate the study

Exclusion Criteria:

* Having comorbidities that affects the corneal surface symptoms and signs
* Having limitation in behavior and awareness

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Blurred Vision symptom | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Eye Pain symptom | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Watery Eyes symptom | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Itchiness symptom | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Grittiness symptom | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Sensitivity to Light symptom | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe

SECONDARY OUTCOMES:
Frequency and Severity of Discomfort when Reading | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Discomfort when Watching TV | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Discomfort when Using Computer | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Discomfort when Driving at Night | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Discomfort when Being Outdoors | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe
Frequency and Severity of Discomfort when Being in Air-Conditioned Areas | From enrollment to 7 days after surgery
  All study outcomes are collected using modified OSDI questionnaire answered by patients before surgery, after surgery and 7 days after surgery.
  These outcomes includes the frequency and severity of:
  * Symptoms: Blurred Vision, Eye Pain, Watery Eyes, Itchiness, Grittiness, Sensitivity to Light
  * Impact on daily life activities: Discomfort when Reading, Discomfort when Watching TV, Discomfort when Using Computer, Discomfort when Driving at Night, Discomfort when Being Outdoors, Discomfort when Being in Air-Conditioned Areas
  Frequency: Never, Some of the time, Most of the time, All of the time Severity: None, Mild, Moderate, Severe

CONTACTS AND LOCATIONS:
Locations (1):
- Ba Ria - Vung Tau Eye Hospital, Bà Ria, Ba Ria - Vung Tau, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152